CLINICAL TRIAL: NCT00314743
Title: A Study Evaluating the Efficacy and Safety of the Oral Neurokinin-1 Antagonist, Aprepitant, in Combination With Ondansetron and Dexamethasone in Patients Undergoing Autologous Peripheral Blood Stem Cell Transplantation
Brief Title: Efficacy & Safety of the Oral Neurokinin-1 Antagonist, Aprepitant, in Combo With Ondansetron & Dexamethasone in Patients Undergoing Auto Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-1192; NCT00285272 (obsolete NCT alias)
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Nausea; Vomiting
Keywords: Patients with Non-Hodgkins Lymphoma or Multiple Myeloma
MeSH Terms: conditions — Nausea; Vomiting; Multiple Myeloma | interventions — Ondansetron; Dexamethasone; Aprepitant

ARMS (2):
- Control (No aprepitant) (Active Comparator): Regimen #1 (BEAM; NHL and HL)
  Carmustine 300 mg/m2 IV on day -7 (premedicate with ondansetron 32 mg IV and dexamethasone 20 mg IV)
  Etoposide 100 mg/m2 IV Q 12 hours x 8 doses on days -6 to -3 (premedicate first daily dose ondansetron 32 mg IV and dexamethasone 20 mg IV)
  Cytarabine 100 mg/m2 IV Q 12 hours x 8 doses on days -6 and -3 (no additional premedication)
  Melphalan 140 mg/m2 IV on day -2 (premedicate with ondansetron 32 mg IV and dexamethasone 20 mg IV)
  Regimen #2 (MM and Amyloidosis)
  Melphalan 100 mg/m2 IV on days -3 and -2 (premedicate each dose with ondansetron 32 mg IV and dexamethasone 20 mg IV)
  Interventions: Drug: Ondansetron; Drug: Dexamethasone
- Experimental (with aprepitant) (Experimental): Aprepitant 125 mg PO will be given 30 minutes prior to the first dose of chemotherapy followed by Aprepitant 80 mg PO QD for the remainder of chemotherapy and continuing for a total of 2 days after completing the regimen.
  Regimen #1 (BEAM; NHL and HL)
  Carmustine 300 mg/m2 IV on day -7 (premedicate with ondansetron 32 mg IV and dexamethasone 10 mg IV)
  Etoposide 100 mg/m2 IV Q 12 hours x 8 doses on days -6 to -3 (premedicate first daily dose ondansetron 32 mg IV and dexamethasone 10 mg IV)
  Cytarabine 100 mg/m2 IV Q 12 hours x 8 doses on days -6 and -3 (no additional premedication)
  Melphalan 140 mg/m2 IV on day -2 (premedicate with ondansetron 32 mg IV and dexamethasone 10 mg IV)
  Regimen #2 (MM and Amyloidosis)
  Melphalan 100 mg/m2 IV on days -3 and -2 (premedicate each dose with ondansetron 32 mg IV and dexamethasone 10 mg IV)
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Aprepitant

INTERVENTIONS:
Drug: Ondansetron
  Other Names: Zofran
Drug: Dexamethasone
Drug: Aprepitant
  Other Names: Emend
  Arms: Experimental (with aprepitant)

SUMMARY:
The purpose of this study is to determine the efficacy of aprepitant in preventing acute and delayed chemotherapy induced nausea and vomiting when administered in combination with intravenous or oral ondansetron and intravenous or oral dexamethasone in the autologous transplant setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Patients deemed eligible to undergo autologous bone marrow or peripheral stem cell transplant therapy per usual transplant inclusion and exclusion criteria
* Patients with Non-Hodgkins Lymphoma, Hodgkins Lymphoma or Multiple Myeloma or Amyloidosis
* Written informed consent

Exclusion Criteria:

* Nausea at baseline
* Chronic use of other antiemetic agent(s)
* Gastrointestinal obstruction or active peptic ulcer
* Radiation therapy to pelvis or abdomen within 1 week before or after study day 1
* Allogeneic stem cell transplant recipient
* Aspartate transaminase (AST) > 3x upper limit of normal (ULN)
* Alanine transaminase (ALT) > 3x ULN
* Bilirubin > 3x ULN
* Alkaline phosphatase > 3x ULN
* Creatinine > 2
* Documented hypersensitivity to any component of study regimen
* Pregnant or lactating women
* Participating in a clinical trial which involves other investigational agent(s)
* Patients taking any of the following medications at time of study day 1: warfarin, oral contraceptives (except for the administration of stopping menses), tolbutamide, phenytoin, midazolam, ketoconazole, rifampin, paroxetine, and/or diltiazem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of aprepitant in preventing acute & delayed chemotherapy induced nausea & vomiting when administered in combination with intravenous or oral ondansetron & intravenous or oral dexamethasone in the autologous transplant setting. | Day 30

SECONDARY OUTCOMES:
To measure the the severity, frequency, and duration of chemotherapy induced nausea and vomiting in patients receiving aprepitant and compare these results to a control group, not receiving aprepitant. | Day 30
To measure the need for breakthrough antiemetics in patients receiving aprepitant and compare these results to the control group | Day 30
To assess the incidence of complications associated with chemotherapy induced nausea and vomiting in patients receiving aprepitant and compare these results to the control group. | Day 30
To assess the safety of aprepitant in combination with ondansetron and dexamethasone in the autologous transplant setting. | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: John F DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu